CLINICAL TRIAL: NCT06337968
Title: Circum-Psoas Block for Arthroscopic Hip Surgery: a Randomized Trial
Brief Title: CPB for Arthroscopic Hip Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Circum-Psoas Block LN
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Acute Pain; Opioid Use
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided circum-psoas block (Active Comparator): Injection of 20ml 0.2% ropivacaine around the antero-lateral margin of psoas major muscle at the level of iliac crest with an in-plane approach under ultrasound guidance. Then the transducer was placed at the level of Lumbar vertebra 5 to obtain the paramedian transverse plane of the intertransverse ligament and lumbosacral ligament. An additional 20ml 0.2% ropivacaine was injected when the needle punctured the lumbosacral ligament.
  Interventions: Procedure: Circum-psoas Block
- Sham block (Placebo Comparator): Perform ultrasound scanning without puncture.
  Interventions: Procedure: Sham block

INTERVENTIONS:
Procedure: Circum-psoas Block — Ultrasound-guided circum-psoas block with 40 mL of treatment drug (Ropivacaine 0.2% [local anesthetic]) 30 minutes prior to induction of anesthesia.
  Arms: Ultrasound guided circum-psoas block
Procedure: Sham block — Perform ultrasound scanning without puncture.
  Arms: Sham block

SUMMARY:
Arthroscopic hip surgery is being increasingly performed to treat both intraarticular and extraarticular hip diseases. Despite the minimally invasive approach, patients undergoing arthroscopic hip surgery still suffer severe pain due to the complex nature of hip innervation. Postoperative pain reduces patient satisfaction and delay patient recovery and discharge. The efficacy of regional anesthesia techniques in postoperative pain management have been proved in various surgeries. However, it remains controversial whether or not peripheral nerve blocks can significantly improve postoperative analgesia after hip arthroscopy.

Several studies have shown that the fascia iliac block cannot improve postoperative analgesia for hip arthroscopy because it blocks only some branches of the lumbar plexus but not the sacral plexus. Circum-Psoas Block (CPB) which has been defined in recent years is able to block the lumbar plexus nerves as well as sacral plexus such as the sciatic, superior gluteal, and inferior gluteal nerves. Therefore, the investigators predict that it can provide effective postoperative analgesia for hip arthroscopy. In this study, the researchers aim to investigate the effectiveness of CPB in hip arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral ambulatory hip arthroscopy
* Age 18 to 70 years
* ASA physical status I to III
* Ability to follow the protocol.

Exclusion Criteria:

* Age <18 or >70 years of age
* BMI above 40
* Contraindications to peripheral nerve blockade
* Pregnancy
* Chronic pain condition requiring opioid intake at home
* Allergy to opioids or local anesthetics
* Patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
pain severity at 6 hours postoperatively | 6 hours postoperatively
  Postoperative pain assessed with NRS pain score (NRS 0: no pain 10: pain as bad as can be) at 1, 6, 12, 24 hours postoperatively. However, to be more precise in our assessment, the effectiveness of each intervention was defined as a reduction in the pain at 6 hours postoperatively.

SECONDARY OUTCOMES:
Postoperative opioid consumption | up to the first 24 hours postoperatively
  Cumulative 24-hr postoperative opioid consumption
Postoperative nausea and vomiting | up to the first 24 hours postoperatively
  Nausea and vomiting intensity score measured by numeric rank score (0:no nausea and no vomiting, 1: have nausea, no vomiting, 2: once vomiting, 3: two or more vomiting).
neurologic evaluation | 1, 6, 24 hours postoperatively
  The dermatomal coverage of sensory block was evaluated by using a cool roller at 1, 6, 24 hours post-surgery. Motor strength was assessed by the following criteria (0: none; 1: muscle flicker without movement; 2: movement, but not against gravity; 3: movement against gravity; 4: movement against some resistance; 5: normal strength).
Patient satisfaction | at the end of 24 hours postoperatively
  Patient satisfaction measured using a numeric rating scale 0 to 10 (0 = unsatisfied; 10 =very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Doctor, Study Director — The Second Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garner M, Alshameeri Z, Sardesai A, Khanduja V. A Prospective Randomized Controlled Trial Comparing the Efficacy of Fascia Iliaca Compartment Block Versus Local Anesthetic Infiltration After Hip Arthroscopic Surgery. Arthroscopy. 2017 Jan;33(1):125-132. doi: 10.1016/j.arthro.2016.10.010. PMID 28003068
- [Background] Baker JF, McGuire CM, Byrne DP, Hunter K, Eustace N, Mulhall KJ. Analgesic control after hip arthroscopy: a randomised, double-blinded trial comparing portal with intra-articular infiltration of bupivacaine. Hip Int. 2011 May-Jun;21(3):373-7. doi: 10.5301/HIP.2011.8390. Epub 2011 Jun 7. PMID 21698591
- [Background] Zheng J, Mi Y, Liang J, Li H, Shao P, Wen H, Wang Y. Circum-Psoas Block versus Supra-Inguinal Fascia Iliaca Block for Postoperative Analgesia in Patients Undergoing Total Hip Arthroplasty: A Randomized Clinical Trial. J Pain Res. 2023 Nov 20;16:3961-3970. doi: 10.2147/JPR.S435159. eCollection 2023. PMID 38026457